CLINICAL TRIAL: NCT06056921
Title: Clinical Study of CD19 Targeting Chimeric Antigen Receptor T Lymphocytes (CAR-T) in the Treatment of Refractory Autoimmune Diseases
Brief Title: Safety and Efficacy of CD19 Targeted CAR-T Therapy for Refractory Autoimmune Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC054
Record Dates: First submitted 2023-08-18; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-08

CONDITIONS: SLE (Systemic Lupus); Sjogren's Syndrome; Systemic Scleroderma; Dermatomyositis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis
Keywords: CAR-T; CD19
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Sjogren's Syndrome; Scleroderma, Systemic; Dermatomyositis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-targeted CAR-T (Experimental): CD19 targeted CAR-T cells treat
  Interventions: Biological: CD19 targeted CAR-T cells

INTERVENTIONS:
Biological: CD19 targeted CAR-T cells — A single infusion of CD19 CAR-T cells will be administered intravenously

SUMMARY:
This is a single arm study to evaluate the efficacy and safety of CD19 targeted CAR-T cells therapy for patients with Refractory Autoimmune Disease

DETAILED DESCRIPTION:
the CD19 targeted CAR-T cell therapies have gained significant results in patients with relapsed and refractory B-cell Leukemia and Lymphoma. Otherwise, some studies have shown that the use of CD19-targeted CAR-T therapy in refractory SLE can improve the autoimmune symptoms of patients, and at the same time, immunosuppressants and hormones can be stopped to maintain long-term autoimmune indicators normal.To verify the safety and efficacy, the investigators launch such a clinical trial using CD19 targeted CAR-T cells for patients with Refractory Autoimmune Disease.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, male or female;
2. diagnosed with one of the following diseases:

   * Systemic Lupus Erythematosus (SLE), EULAR/ACR 2019 standard;
   * Sjogren's Syndrome (SS), 2016 ACR/EULAR standard;
   * Systemic Scleroderma (SSc), 2013 ACR/EULAR Standards;
   * Dermatomyositis (DM), 2017 EULAR/ACR classification standard + one positive myositis specific antibody (Jo-1, Zo, EJ, PL-7, KS, OJ, PL-12, YRS, Anti-NXP-2, Anti-TIF1g, Anti-Mi-2, Anti-SAE, Anti-MDA-5, Anti-SRP, Anti-HMGCR);
   * Anti-neutrophil cytoplasmic antibody associated vasculitis (ANCA-AAV), including granulomatosis with polyangiitis (GPA), or microscopic vasculitis (MPA), or eosinophilic granulomatosis with polyangiitis (EGPA), 2022 ACR/EULAR standard.
3. Disease activity meets the following requirements:

   * SLEDAI score ≥8 for SLE patients;
   * For SS patients, ESSDAI≥14 points;
   * For patients with SSc, mRSS score in the range of 10-35 (including the boundary value) with interstitial pneumonia (ILD);
   * Patients with DM who have been diagnosed for at least 1 year and meet the following conditions:

     1. Skin rash VAS score (based on MDAAT) ≥3cm with at least 3 abnormalities in CSM;

     2, muscle biopsy pathology or muscle nuclear magnetic evidence of active inflammation;

     3. Bilateral manual muscle strength test (MMT-8) is less than 125/150, and at least 2 additional Core set measures (CSM) meet the following criteria: Patient score, 10 cm visual analogue scale (VAS) no less than 2.0 cm; b. Physician score, no less than 2.0 cm on the 10 cm VAS scale; c. Health Assessment Questionnaire (HAQ) disability index (Appendix 10) of not less than 0.25; d. Elevation of at least one muscular enzyme (including creatine kinase (CK), aldolase, lactate dehydrogenase (LDH), alanine aminotransferase (ALT) and aspartate aminotransferase (AST)), with a minimum level of 1.3× the upper limit of normal; e. Disease activity score of extramuscular organs, no less than 1.0 cm on the 10 cm VAS scale (this VAS is the physician's comprehensive assessment of myositis disease Activity Assessment Tool (MDAAT) based on the general condition, skin, bone, gastrointestinal, lung, and heart scale activity score);
   * For ANCA-AAV patients, the BVAS score was ≥15.
4. ECOG 0~1 score;
5. The functions of important organs are basically normal:

   * Hematology: hemoglobin ≥60g/L, platelet count ≥30×109/L;
   * Cardiac function: Left ventricular ejection fraction (LVEF) ≥55%, no obvious abnormality in electrocardiogram;
   * Renal function: eGFR≥30ML/min/1.73m2;
   * Liver function: AST and ALT≤3.0 ULN, total bilirubin ≤2.0 ULN;
   * Lung function: DLCO≥40% predicted value; FVC≥50% expected value;
   * Have criteria for simple or intravenous blood collection, and no other contraindications for cell collection;
6. The subject of childbearing age has a negative urine pregnancy test result and agrees to take effective contraceptive measures during the test period until 1 year after the infusion;
7. The patient or his/her guardian agrees to participate in the clinical trial and signs the informed consent, indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study.

Exclusion Criteria:

1. Had previously received CAR T cell therapy;
2. patients with serious heart, liver, lung, blood system, endocrine system diseases, and the risk of participating in the trial is higher than the benefit judged by the researcher;
3. There is an active or uncontrollable infection that requires systemic treatment within 1 week prior to screening;
4. have previously received hematopoietic stem cell transplantation or solid organ transplantation (except corneal and hair transplantation), or have grade 2 or higher acute graft-versus-host disease (GVHD) within 2 weeks prior to screening;
5. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal reference value range; Or hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal reference value range; Or positive for human immunodeficiency virus (HIV) antibodies; Or syphilis test positive; Or cytomegalovirus (CMV) DNA test positive;
6. Had received live vaccine within 4 weeks before screening;
7. pregnancy test positive;
8. Patients with malignant diseases such as malignant tumors before screening, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery;
9. Patients who had participated in other clinical trials within 3 months prior to screening;
10. Situations in which other investigators consider it inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after CD19 CAR-T cells infusion [Safety and Tolerability] | 1 month
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
Obtain the maximum tolerated dose of CD19 CAR-T cells[Safety and Tolerability] | 1month
  Dose-limiting toxicity after cell infusion
Efficacy of CAR-T cell preparations in Refractory systemic lupus erythematosus [Effectiveness] | 3 months
  The efficacy is assessed by SRI-4 response rate at 3M，SRI-4 response rate at 3M means Percentage of patients who met all three of the following conditions at 3M after refusion:
  1. The SLEDAI-2K rating dropped by at least 4 points
  2. No deterioration in PGA scores on a 3-point scale (deterioration is defined as an increase of ≥0.3 points from baseline score)
  3. No new manifestations of organ system involvement (new system involvement is defined as one or more new symptoms of BILAG grade A or two or more symptoms of BILAG B)
Efficacy of CAR-T cell preparations in Refractory Systemic scleroderma [Effectiveness] | 3 months
  The efficacy is assessed by Change value of The EULAR Sjögren's syndrome disease activity index（ESSDAI）score at 3M
Efficacy of CAR-T cell preparations in Refractory Sjogren's syndrome [Effectiveness] | 3 months
  The efficacy is assessed by Change value of modified Rondan skin score（mRSS） at 3M； The evaluator palpated 17 areas of the patient's body. The skin thickness of each area was calculated on a scale of 0 to 3 points. The total score was 51 points, 0 was normal skin with fine lines and no skin thickening. 1 is divided into mild skin thickening, the inspector can easily use two fingers to pinch the skin to form wrinkles, skin fine lines can also exist; 2: moderate skin thickening, more difficult to pinch the skin to form wrinkles, skin fine lines disappear; 3 is classified as severe skin thickening, unable to pinch the skin to form wrinkles.
Efficacy of CAR-T cell preparations in Refractory dermatomyositis [Effectiveness] | 3 months
  The efficacy is assessed by CSM Total Improvement Score (TIS) 20/40/60 improvement rate at 3M；3M CSM Total Improvement Score (TIS) 20/40/60 Improvement rate: defined as the proportion of patients with a TIS score of 20-40,40-60, and ≥60 at 3M posttransfusion
Efficacy of CAR-T cell preparations in Refractory The antineutrophil cytoplasmic antibody-associated vasculitides [Effectiveness] | 3 months
  The efficacy is assessed by response rate at 3M； Defined as the percentage of patients whose BVAS score decreased to 0 at 3M after reinfusion in the absence of glucocorticoids and other therapeutic agents

SECONDARY OUTCOMES:
AUCS of CD19 CAR-T cells [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 90 days
CMAX of CD19 CAR-T cells [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of CD70 CAR-T cells expanded in peripheral blood
TMAX of CD19 CAR-T cells[Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
Pharmacodynamics of CD19 CAR-T cells[Cell dynamics] | 3 months
  Pharmacodynamics is defined as the degree of B cell clearance at each time point
Immunogenicity after infusion of CD19 CAR-T | 2 years
  Positive rate of anti-CAR antibody in peripheral blood
Immunological reconstitution of CAR-T after infusion of CD19 CAR-T | 2 years
  The change curve of B cells in peripheral blood after transfusion;

OTHER OUTCOMES:
Refractory systemic lupus erythematosus -specific secondary study endpoint [Effectiveness] | 2 years
  SLEDAI-2K change curve within 2 years after the transfusion or subjects withdrew from the study for various reasons (whichever happened first);
Refractory Systemic scleroderma-specific secondary study endpoint [Effectiveness] | 2 years
  ESSDAI change curve within 2 years after transfusion or subjects withdrew from the study for various reasons (whichever happened first); ESSPRI change curve;
Refractory Sjogren's syndrome-specific secondary study endpoint [Effectiveness] | 2 years
  DLCO change curve within 2 years after transfusion or subjects withdrew from the study for various reasons (whichever happened first);
Refractory dermatomyositis-specific secondary study endpoint [Effectiveness] | 2 years
  3M CDASI score changes (Appendix 14); CDASI score change curve within 2 years after transfusion or subjects withdrew from the study for various reasons (whichever happened first);
Refractory The antineutrophil cytoplasmic antibody-associated vasculitides -specific secondary study endpoint [Effectiveness] | 2 years
  BVAS score within 2 years after retransfusion or when subjects withdrew from the study for various reasons (whichever occurred first).

CONTACTS AND LOCATIONS:
Overall Officials: Liyun Zhang, M.D, Principal Investigator — Shanxi Bethune Hospital
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China